CLINICAL TRIAL: NCT07265479
Title: A Randomized, Double-Blind, Vehicle-Controlled (Period 1) and Open-Label (Period 2) Phase 3 Study to Investigate the Safety and Efficacy of Tapinarof Cream, 1% in Pediatric Participants Ages 3 Months to < 24 Months With Atopic Dermatitis
Brief Title: A Study to Investigate Safety and Efficacy of Tapinarof Cream, 1% in Participants Ages 3 Months to < 24 Months With Atopic Dermatitis
Acronym: Adoring
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OG0505-3104
Record Dates: First submitted 2025-11-21; First posted 2025-12-04 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-11

CONDITIONS: Atopic Dermatitis
Keywords: Pediatric Atopic Dermatitis; Eczema; tapinarof; topical
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — tapinarof

STUDY DESIGN:
Intervention Model Description: Following a screening period of up to 30 days, eligible participants will be randomly assigned to one of two groups for up to 8 weeks. During this time-called the Double-Blind Period-2 out of 3 participants will receive the active treatment (tapinarof cream, 1%), while 1 out of 3 will receive a vehicle cream (placebo).
  Following completion of the Double-blind period, participants will enter the 48-week Open Label Period and will be treated as needed.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tapinarof cream (Experimental): Tapinarof cream, 1%, applied topically once daily
  Interventions: Drug: Tapinarof cream, 1%
- Vehicle cream (Placebo Comparator): Vehicle cream is applied topically once daily for up to 8-weeks.
  Interventions: Drug: Vehicle Cream

INTERVENTIONS:
Drug: Tapinarof cream, 1% — Tapinarof cream, 1%: Applied topically once daily to lesions on participant's skin during the Double-Blind period. During the Open-Label Period, it will be applied once daily to lesions, as needed.
  Other Names: OG-0505; DMVT-505; GSK2894512A; GSK28994512; STI-1001; WBI-1001
  Arms: Tapinarof cream
Drug: Vehicle Cream — Applied topically once daily to lesions on participant's skin during the Double-Blind period.
  Arms: Vehicle cream

SUMMARY:
The purpose of this global Phase 3 clinical study is to investigate the safety and efficacy of tapinarof cream, 1% in participants ages 3 months to 23 months (inclusive) with atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Infants and toddlers 3 months to <24 months (post-natal) of age at the Screening visit.
* Clinical diagnosis of atopic dermatitis (AD), AD covering >5% Body Surface Area (BSA) and validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD) score of 2, 3 or 4
* Legal guardian or primary caregiver is willing and able to sign informed consent form before any study-related activities
* Legal guardian or primary caregiver is able and willing to adhere to protocol requirements

Exclusion Criteria:

* Significant neurological disorder or history of seizure
* Clinically significant cardiac rhythm or functional cardiac disorder
* History of sudden infant death in a sibling
* Clinically significant chromosome abnormality
* History of or ongoing serious illness or medical, physical or psychiatric condition(s) that may interfere with the participant's participation
* Diseases that could cause pruritic and/or sleep disruption
* Immunocompromised
* Current chronic or acute infection requiring treatment
* Use of prohibited medication(s) or procedure(s)
* Use of prohibited medications by mother if breastfeeding participant

Ages: 3 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2025-12-29 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who have a validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD) score of clear or almost clear (0 or 1) and a minimum 2-grade Improvement from Baseline to Week 8 | Baseline to last planned visit in the Double-Blind Period, up to 8 weeks.
  The vIGA-AD is a global assessment of the current state of the disease. It is a static 5-point scale used to grade overall disease severity (scalp excluded), as determined by the investigator, using the clinical characteristics of erythema, induration/papulation, lichenification, oozing/crusting. The vIGA-AD ranges from 0 to 4 and is reported as Clear (0), Almost clear (1), Mild (2), Moderate (3), and Severe (4). Higher vIGA-AD scores represent more severe disease.
Percentage of participants who enter with or achieve have a validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD) score of clear or almost clear (0 or 1) and a minimum 2-grade Improvement at least once during the Open-Label Period | Baseline to the end of the Open-Label Period, up to 56 weeks.
  The vIGA-AD is a clinical tool for assessing the current state/severity of a subject's atopic dermatitis at a given timepoint.. It is a static 5-point scale used to grade overall disease severity (scalp excluded), as determined by the investigator, using the clinical characteristics of erythema, induration/papulation, lichenification, oozing/crusting. The vIGA-AD ranges from 0 to 4 and is reported as Clear (0), Almost clear (1), Mild (2), Moderate (3), and Severe (4). Higher vIGA-AD scores represent more severe disease.

SECONDARY OUTCOMES:
Percentage of participants with ≥ 75% improvement in Eczema Area and Severity Index (EASI) Score from Baseline to Week 8. | Baseline to last planned visit in the Double-Blind Period, up to 8 weeks.
  The EASI is a scoring system that takes into account the overall severity of disease based on lesion severity and the %BSA affected with atopic dermatitis. The EASI is a composite score ranging from 0 -72 that takes into account the degree of erythema, edema/papulation, excoriation, and lichenification (each scored from 0 to 3 separately) for each of four body regions, with adjustment for the %BSA involved for each body region relative to the whole body. The subject's scalp is excluded from this assessment. A higher EASI score represents more severe disease.
Mean change in percentage of total body surface area (%BSA) affected from Baseline to Week 8 | Baseline to last planned visit in the Double-Blind Period, up to 8 weeks.
  Assessment of %BSA is an estimate of the percentage of total involved skin with atopic dermatitis. Estimates were made using the handprint method, where the full palmar hand of the participant (fully extended palm, fingers and thumbs together) represented approximately 1% of the total BSA. Body regions are assigned a specific number of handprints with associated percentages (Head and neck = 10% [10 handprints], upper extremities = 20% [20 handprints], trunk (including axillae and groin) = 30% [30 handprints], lower extremities, including buttocks, = 40% [40 handprints]). Estimates of the percent involvement of each body region will be multiplied by the fraction of total body area to obtain the total %BSA involved by region and overall.
Percentage of participants with ≥ 90% improvement in Eczema Area and Severity Index (EASI) score from Baseline to Week 8 | Baseline to last planned visit in the Double-Blind Period, up to 8 weeks.
  Severity Index (EASI) score from Baseline to Week 8 Description: The EASI is a scoring system that takes into account the overall severity of disease based on lesion severity and the extent of percent body surface area affected with atopic dermatitis. The EASI is a composite score ranging from 0 -72 that takes into account the degree of erythema, edema/papulation, excoriation, and lichenification (each scored from 0 to 3 separately) for each of four body regions, with adjustment for the percent body surface area involved for each body region relative to the whole body. A higher EASI score represents more severe disease.
Number of participants with one or more Treatment Emergent Adverse Events (TEAEs) | Baseline to last planned visit in the Double-Blind Period, up to 8 weeks
  TEAEs are AEs that started on or after the first dose of study medication.
Number of participants with one or more Treatment Emergent Adverse Events (TEAEs) | Baseline to the end of the Open-Label Period, up to 56 weeks
  TEAEs are AEs that started on or after the first dose of study medication.
Percentage of participants with one or more Treatment Emergent Adverse Events (TEAEs) | Baseline to last planned visit in the Double-Blind Period, up to 8 weeks .
  TEAEs are AEs that started on or after the first dose of study medication.
Percentage of participants with one or more Treatment Emergent Adverse Events (TEAEs) | Baseline to the end of the Open-Label Period, up to 56 weeks.
  TEAEs are AEs that started on or after the first dose of study medication.
Investigator-assessed Local Tolerability Scale (LTS) scores by visit (overall) | Baseline to last planned visit in the Double-Blind Period, up to 8 weeks
  The LTS measures the presence and overall degree of irritation at the application site(s) using a 5-point scale, where 0 indicates no irritation and 4 very severe irritation.
Investigator-assessed Local Tolerability Scale (LTS) scores by visit (overall) | Beginning of Open-Label to the end of the Open-Label Period, up to 48 weeks.
  The LTS measures the presence and overall degree of irritation at the application site(s) using a 5-point scale, where 0 indicates no irritation and 4 very severe irritation.
Investigator-assessed Local Tolerability Scale (LTS) scores by visit (sensitive areas) | Baseline to last planned visit in the Double-Blind Period, up to 8 weeks
  The LTS measures the presence and overall degree of irritation at the application site(s) using a 5-point scale, where 0 indicates no irritation and 4 very severe irritation.
Investigator-assessed Local Tolerability Scale (LTS) scores by visit (sensitive areas) | Beginning of Open-Label to the end of the Open-Label Period, up to 48 weeks.
  The LTS measures the presence and overall degree of irritation at the application site(s) using a 5-point scale, where 0 indicates no irritation and 4 very severe irritation.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Lead Late-Stage Clinical Development, Study Director — Organon and Co
Locations (49):
- United States (39):
  - AllerVie Clinical Research, Birmingham, Alabama
  - Dermatology Trial Associates, Bryant, Arkansas
  - Dermatology Research Associates, Los Angeles, California
  - Integrative Skin Science and Research, Sacramento, California
  - Allergy and Asthma Medical Group and Research Center, San Diego, California
  - Clinical Trials Research Institute, Thousand Oaks, California
  - Clarity Dermatology, Castle Rock, Colorado
  - Skin Care Research, LLC., Boca Raton, Florida
  - APEX Clinical Trials, Jacksonville, Florida
  - TruDerm Research, Wellington, Florida
  - Dermatology Affiliates Research Institute, Atlanta, Georgia
  - Cleaver Medical Group Dermatology, Inc, Cumming, Georgia
  - Ada West Research, Meridian, Idaho
  - Northwestern University, Chicago, Illinois
  - Endeavor Health Clinical Operations, Skokie, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - The Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - Equity Medical, LLC, Bowling Green, Kentucky
  - Lawrence J Green, MD LLC, Rockville, Maryland
  - Oakland Hills Dermatology P.C, Auburn Hills, Michigan
  - Minnesota Clinical Study Center, New Brighton, Minnesota
  - SKY Integrative Medical Center, Ridgeland, Mississippi
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Skin Cancer and Dermatology Institute, Reno, Nevada
  - Forest Hills Dermatology Group, Kew Gardens, New York
  - Bobby Buka MD, PC, New York, New York
  - Equity Medical, LLC, The Bronx, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Wright State Physicians, Fairborn, Ohio
  - Allergy Asthma and Clinical Research Center, Oklahoma City, Oklahoma
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - National Allergy and Asthma Research, LLC., North Charleston, South Carolina
  - The University of Texas Health Science Center at Houston, Bellaire, Texas
  - Dermatology Treatment and Research Center, Dallas, Texas
  - Stryde Consulting, LLC, Southlake, Texas
  - Dermatology Specialists of Spokane, Spokane, Washington
- Canada (10):
  - Dermatology Research Institute, Calgary, Alberta
  - CARe Clinic (Central Alberta Research Clinic), Red Deer, Alberta
  - Dr. Chih-ho Hong Medical Inc., Surrey, British Columbia
  - Manitoba Allergy Research Inc., Winnipeg, Manitoba
  - Maritime Dermatology, Halifax, Nova Scotia
  - Halton Pediatric Allergy, Burlington, Ontario
  - Triple A Lab Inc., Hamilton, Ontario
  - Allergy Research Canada Inc., Niagara Falls, Ontario
  - Origins Dermatology Centre, Regina, Saskatchewan
  - Skinsense Medical Research, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No